CLINICAL TRIAL: NCT05034393
Title: Real-World Data on First-line Treatment of Hormone Receptor-positive, HER2-negative, Metastatic Breast Cancer in Brazil
Acronym: BRAVE
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Brazilian Breast Cancer Study Group (GBECAM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: LACOG 0221
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with de novo or recurrent HR-positive HER2-negative mBC: Patients diagnosed with de novo or recurrent HR-positive HER2-negative mBC from January 2018 to December 2020

SUMMARY:
This study aims to describe in detail the patient journey from diagnosis to the beginning of treatment and patterns of care of hormone receptor- positive, HER2-negative de novo or recurrent metastatic breast cancer between January 2018 and December 2020 in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old
* Histologically confirmed hormone receptor-positive HER2-negative invasive breast cancer
* Hormone receptor-positive defined as 1% to 100% of tumor nuclei positive for Estrogen - - Receptor and/or Progesterone Receptor, as per ASCO/CAP Guideline 2020 - or Allred score of ≥3
* HER2-negative defined as IHC result is 0/1+ or 2+ with ISH negative as per ASCO/CAP Guideline 2018
* Diagnosed with de novo or recurrent metastatic breast cancer between January 2018 -and December 2020
* Public health system or private health system

Exclusion Criteria:

* Male Breast Cancer
* First-line treatment for mBC received through clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women histologically confirmed hormone receptor-positive HER2-negative invasive breast cancer
Study Population: The study will be performed in up to 15 sites in Brazil so that the recruitment target is reached within defined milestones. An adequate geographical distribution of sites within Brazil will be pursued to strengthen representation of Brazilian population. Considering the incidence of mBC.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
The proportion of type of first-line treatment | from January 2018 to December 2020

SECONDARY OUTCOMES:
The PFS, defined as time from treatment start until progression (by image or physical exam) or death | from January 2018 to December 2020
First-line treatment according to the drug name by type of health care coverage (public vs private) | from January 2018 to December 2020
The PFS will be evaluated by type of health care coverage (public vs private). | from January 2018 to December 2020
Timeline from first symptom to diagnosis | from January 2018 to December 2020
Timeline from diagnosis to molecular test | from January 2018 to December 2020
Timeline from diagnosis to the beginning of treatment | from January 2018 to December 2020
Patients' socioeconomic characteristics | from January 2018 to December 2020
Patients' demographics characteristics | from January 2018 to December 2020
BC pathological characterization | from January 2018 to December 2020
Rate of diagnostic tests to define breast cancer molecular subtypes performed | from January 2018 to December 2020

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, Principal Investigator — Latin American Cooperative Oncology Group
Locations (15):
- Brazil (15):
  - CINPAM - Centro Integrado de Pesquisa da Amazônia, Manaus, Amazonas
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - CLION - Clínica de Oncologia (Oncoclínicas), Salvador, Estado de Bahia
  - Hospital Sírio-Libanês DF, Brasília, Federal District
  - IGESDF - Instituto de Gestão Estratégica em Saúde do Distrito Federal, Brasília, Federal District
  - Instituto do Câncer Brasil - Unidade Pantanal, Corumbá, Mato Grosso do Sul
  - Instituto do Câncer Brasil - Unidade Três Lagoas, Três Lagoas, Mato Grosso do Sul
  - Instituto de Hematologia e Oncologia Curitiba (Oncoclínicas), Curitiba, Paraná
  - CPO - Centro Paraibano de Oncologia (Oncoclínicas), João Pessoa, Paraíba
  - HINJA - Hospital Jardim Armália, Volta Redonda, Rio de Janeiro
  - CEPESG - Centro de Pesquisa e Educação da Serra Gaúcha, Caxias do Sul, Rio Grande do Sul
  - HMV - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto do Câncer Brasil - Unidade Andradina, Andradina, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided